CLINICAL TRIAL: NCT05995158
Title: Metagenomic Analysis of the Link Between Periodontitis and Smoking: Case-control Study
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Jazia Alblowi, Associate Professor, King Abdulaziz University
Other Study IDs: 127-10-18
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Condition, Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples of the subgingival plaque
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers ≥ 10 cigarettes/day: metagenomic testing of the subgingival plaque samples 16S rRNA metagenomic testing (sampling, extraction and sequencing of the oral microbiome in the samples)
  Interventions: Procedure: Metagenomic testing of the subgingival plaque samples
- Smokers < 10 cigarettes/day: metagenomic testing of the subgingival plaque samples 16S rRNA metagenomic testing (sampling, extraction and sequencing of the oral microbiome in the samples)
  Interventions: Procedure: Metagenomic testing of the subgingival plaque samples
- non-smokers: metagenomic testing of the subgingival plaque samples 16S rRNA metagenomic testing (sampling, extraction and sequencing of the oral microbiome in the samples)
  Interventions: Procedure: Metagenomic testing of the subgingival plaque samples

INTERVENTIONS:
Procedure: Metagenomic testing of the subgingival plaque samples — sampling, extraction and sequencing of the oral microbiome in the samples

SUMMARY:
Periodontitis is a widely prevalent disease worldwide that has serious public health consequences. Its prognosis includes tooth loss and edentulism, a condition that negatively affects chewing causing functional disability; and esthetics causing social impairment. Consequently, periodontitis may end up causing marked impairment of the quality of life of the affected patients, impairment of general health and increasing the dental care costs significantly.

Dysbiotic changes in the oral microbiome arise after some microbial species are enriched by primary products resulting from tissue breakdown due to gingivitis. It then triggers the host cells to produce proteinases that mediate loss of marginal periodontal ligaments, apical migration of the junctional epithelium and apical spread of bacterial biofilm.

However, the dysbiotic changes may be more likely to occur in some patients rather than others due to certain risk factors including smoking and immuneinflammatory responses. Thus, the severity of periodontal disease in these patients would be higher. Tobacco smoking is no longer considered to be a habit, but a dependence to nicotine and a chronic relapsing medical disorder. Among its detrimental effects on general health, tobacco smoking increases the risk of periodontitis by 2 to 5 folds. This takes place by increasing the dysbiotic changes in the oral microbiome and so, increasing the severity and extent of the periodontal disease at a younger age. Therefore, smoking has been considered as a modifying factor of periodontitis that should be considered upon periodontitis case grading definition.

Therefore, this research aims to identify the difference in dysbiosis between the three categories of periodontitis, trying to understand the cause of the resistance of each category to treatment compared to the milder category.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Patients with periodontitis.
* Probing pocket depth ≥ 4 mm.
* Teeth with CAL≥ 3 mm at ≥2 non-adjacent teeth.
* Clinical indication and/or patient request for treatment of the periodontal condition.

Exclusion Criteria:

* Patients with any systemic diseases.
* Pregnant females.
* Patients who took any antibiotic in the past month.
* Handicapped and mentally retarded patients.
* Patients undergoing radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients clinically diagnosed to have chronic periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
oral microbiome composition by NGS sequencing using next generation sequencer | 1 month

SECONDARY OUTCOMES:
Probing depth (mm) by periodontal probe | 1 month
Bleeding on probing tested by a periodontal probe % of sites with bleeding on probing | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jazia A Alblowi, PhD, Principal Investigator — King Abdulaziz University Faculty of Dentistry
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No